CLINICAL TRIAL: NCT05757557
Title: Perioperative Nitric oxiDE-conditioning, Produced by Plasma-chemical Synthesis Technology, For prevEnt Acute kidNey Injury During carDiac surgEry in Patients With chRonic Kidney Disease (DEFENDER-trial)
Brief Title: Perioperative Nitric Oxide Prevents Acute Kidney Injury in Cardiac Surgery Patients With Chronic Kidney Disease
Acronym: DEFENDER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Nikolay Kamenshchikov, MD, PhD, Head of Laboratory, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DEFENDER
Record Dates: First submitted 2023-02-11; First posted 2023-03-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Disease; Chronic Kidney Disease; Cardiac Surgery; Cardiopulmonary Bypass
Keywords: Acute Kidney Disease; Nitric Oxide; Chronic Kidney Disease; Cardiopulmonary Bypass; Cardiac Surgery; Prevention
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Oxygen-air mixture without NO after intubation, during CPB, and six hours after surgery.
  Interventions: Drug: Sham treatment
- 80-ppm NO (Experimental): NO will be supplemented at 80-ppm concentration to cardiac surgery patients perioperative after trachea intubation, during CPB, and six hours after surgery.
  Interventions: Drug: 80-ppm NO

INTERVENTIONS:
Drug: Sham treatment — Sham treatment: Oxygen-air mixture without NO after intubation, during CPB, and for six hours after surgery.
  Other Names: Oxygen-Air Mixture
  Arms: Control group
Drug: 80-ppm NO — NO will be supplemented at 80-ppm concentration to cardiac surgery patients perioperatively after trachea intubation, during CPB, and for six hours after surgery.
  Other Names: Nitric Oxide
  Arms: 80-ppm NO

SUMMARY:
The protective nitric oxide (NO) effects are mediated by selective pulmonary vasodilation and improvement of arterial oxygenation in hypoxemic patients by reducing intrapulmonary shunting and improving ventilation-perfusion coordination. Inhaled NO has been used for years to treat acute respiratory failure and pulmonary hypertension in anesthesia and intensive care. The nephroprotective role of NO was studied in an experimental model of contrast-induced nephropathy. The primary aim of this prospective, double-blind, randomized, parallel-group, controlled trial is to test the hypothesis that perioperative conditioning of patients with NO at a dose of 80 ppm, obtained by plasma-chemical synthesis technology, through a ventilator and an extracorporeal circulation circuit reduces the incidence of acute kidney injury (AKI) in patients with an initially high risk of kidney damage due to the presence of preoperative chronic kidney disease (CKD). The study is interventional. Examination and treatment of patients is carried out in accordance with the approved standards of medical care for the relevant diseases. During the study, no experimental or unregistered (not approved for use) medical or diagnostic procedures in the territory of the Russian Federation will be carried out. The study includes patients admitted to the Cardiac Surgery Department of Cardiology Research Institute of Tomsk NRMC for elective surgery with high risk of AKI in the perioperative period

DETAILED DESCRIPTION:
NO abruptly relaxes vascular smooth muscle, leading to pulmonary vasodilation without appreciable hemodynamic effect on extrapulmonary vessels (selective pulmonary vasodilation). In addition, NO expands the smooth muscle of constricted bronchi, which may improve arterial oxygenation in hypoxemic patients by reducing intrapulmonary shunting and improving ventilation-perfusion coordination. NO has been used for many years to treat acute respiratory failure and pulmonary hypertension in anesthesia and intensive care. Several experimental and clinical studies have demonstrated extrapulmonary effects of NO, predominantly on diuresis and natriuresis, platelet function, and modulation of the immune response. The nephroprotective role of NO was studied in an experimental model of contrast-induced nephropathy.

This study is prospective, double-blind, randomized, parallel-group, controlled trial. In regard to medical procedures, this study is interventional. Examination and treatment of patients is carried out in accordance with the approved standards of medical care for the relevant diseases. During this study, no experimental or unregistered (not approved for use) medical or diagnostic procedures in the territory of the Russian Federation is carried out.

The primary aim of the study is to test the hypothesis that perioperative conditioning of patients with NO at a dose of 80 ppm, obtained by plasma-chemical synthesis technology, through a ventilator and an extracorporeal circulation circuit reduces the incidence of AKI in patients with an initially high risk of kidney damage due to the presence of preoperative CKD.

Secondary objectives of the study include the following:

* To test the hypothesis that perioperative conditioning of patients with NO at a dose of 80 ppm, obtained using plasma-chemical synthesis technology, through the ventilator circuit and the extracorporeal circulation circuit is associated with an improvement in regional kidney oximetry.
* To test the hypothesis that the method of monitoring regional kidney oximetry in the para-infrared spectrum is an effective intraoperative method for quantifying the organoprotective effect of NO-therapy.
* To test the hypothesis that perioperative conditioning of patients with NO at a dose of 80 ppm, obtained by plasma-chemical synthesis technology, through the ventilator circuit and the extracorporeal circulation circuit is associated with optimization of endogenous NO homeostasis, determined by the level of NO in the air exhaled by the patient.
* To test the hypothesis that perioperative conditioning of patients with NO at a dose of 80 ppm, obtained using plasma-chemical synthesis technology, through the ventilator circuit and the extracorporeal circulation circuit is associated with an improvement in the global oxygen status of the body, assessed using ΔPCO2/ΔContO2.
* To test the hypotheses that perioperative conditioning of patients with NO at a dose of 80 ppm, obtained using the plasma-chemical synthesis technology through the ventilator circuit and the extracorporeal circulation circuit, reduces the frequency and severity of other organ damage and complications: cardiac, pulmonary, hemorrhagic, neurological, infectious complications, multiple organ failure after surgery, duration of mechanical ventilation, time of stay in the intensive care unit, in-hospital and 30-day mortality in patients with CKD.

Currently, there is no convincing evidence of the benefits or harms of additional NO therapy as part of the anesthesia management of cardiac surgery in patients at high risk of developing AKI. Therefore, there is no reason to believe that randomization into study groups creates additional risks/benefit for patients.

Regardless of the results of randomization, the decision on the relevance of perioperative administration of NO for cardiac surgery in each case is made by a medical consultation, including a cardiac surgeon, an anesthesiologist and a cardiologist immediately after the patient is included in the study.

The study includes patients admitted to the Cardiac Surgery Department of the Research Institute of Cardiology, Tomsk National Research Medical Center for elective surgery, and who have a high risk of AKI in the perioperative period. The frequency of AKI was chosen as the primary endpoint because the manifestation of multiple organ damage in the vast majority of cases begins with renal dysfunction. AKI is a self-perpetuating condition that causes respiratory, cardiac, and cerebral failure.

After patients enter the operating room, they are randomly assigned to the study intervention group (80 ppm NO) or control group. The devices available in the clinic, discussed above, that perform synthesis, supply of inhaled NO, and monitor NO, nitrogen dioxide (NO2) in the supply line directly during therapy, will be used NO. In the NO group, the final concentration of NO is 80 ppm. Patients in the control group will receive a standard NO-free oxygen-air mixture. NO will be supplied immediately after the patient is intubated through the anesthesia machine circuit throughout the operation, followed by the NO delivery through the oxygenator of the cardiopulmonary bypass (CPB) machine throughout the CPB, after weaning from the CPB through the anesthesia machine circuit until the end of the operation and within 6 hours after interventions through the ventilator circuit or through a face mask if the patient will be extubated earlier.

The choice of NO dose and exposure time for clinicians is based on two basic principles:

1. the applied dose of NO and its exposure time are safe for patients;
2. the applied dose of NO and its exposure time are sufficient to provide potential protective effects.

Devices for NO therapy (for the delivery of NO at all stages of the study) are developed at the Research and Production Center for Physics of the Federal State Unitary Enterprise "Russian Federal Nuclear Center - All-Russian Research Institute of Experimental Physics".

For the delivery of nitric oxide at all stages of the study, a device for plasma-chemical synthesis of nitric oxide will be used. For production and for all processes of the product life cycle, the International Certificate of Conformity ISO 13485:2016 Medical Devices - Quality Management Systems, No. GKRU-0072-MD has been received. The device used in this study makes it possible to produce nitric oxide from the air in a gas discharge by generating a repetitively pulsed diffuse discharge excited in an atmospheric pressure air in a gap with a sharply nonuniform electric field. Such a discharge ensures efficient synthesis of nitric oxide in a nonequilibrium low-temperature plasma.

In this study a multimodal approach will be applied to reduce the incidence of acute kidney injury after cardiac surgery. Strategies for optimizing renal outcomes will be applied during the study. Implementation of the Kidney Disease: Improving Global Outcomes guidelines for nephroprotection will be the standard for all patients during the study (Close monitoring of renal function; Functional haemodynamic monitoring; Optimizing fluid status and haemodynamics; Avoidance of hyperglycaemia; Avoidance of radiocontrast and discontinuation of nephrotoxic medications). During CPB, all patients will receive a goal-directed perfusion strategy. In this study it is aimed to maintain a high-normal oxygen delivery target at > 280 ml min m2.

Thus, this study is supposed to assess the potential benefit of perioperative NO conditioning in the era of proven technologies for preventing AKI and determine its potential relevance in the concept of multimodal protection.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with CPB
* Age > 18 years
* Signed informed consent
* CKD (cGFR <60 mL/min/1.73 m2)
* Positive decision of council of physicians on individual safety of perioperative administration of NO

Exclusion Criteria:

* Emergency surgery (including that in ACS)
* cGFR <15 mL/min/1.73 m2
* Administration of potentially nephrotoxic drugs within 24 hours before surgery (radiocontrast agents, antimicrobial therapy with aminoglycosides and / or amphotericin)
* Critical preoperative status (preoperative need for mechanical ventilation, inotropes, circulatory support)
* Pregnancy
* Ongoing enrolment in other randomized clinical trial
* Previous randomization in DEFENDER trial
* Active endocarditis and/or sepsis
* Pulmonary hypertension higher than stage II (systolic pulmonary pressure over 65 mmHg according to data of preoperative transthoracic echocardiography
* Condition after kidney transplantation
* Ongoing AKI caused by glomerulonephritis, interstitial nephritis, renal artery occlusion, or postrenal occlusion
* Cardiac surgery with hypothermic circulatory arrest
* Left ventricular ejection fraction < 30%
* Single kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI (%) | 7 days
  Difference between groups in the incidence of AKI in patients with CKD are assessed as percentage after cardiac surgery according to KDIGO criteria.

SECONDARY OUTCOMES:
Incidence of low cardiac output syndrome (%) | 24 hours
  Difference between groups in the incidence of low cardiac output syndrome (decrease in the incidence of low cardiac output syndrome) with the definition of its type (with dysoxia, without dysoxia, microcirculatory distress). It is a combined point and includes an increase (or various combinations of these parameters according to the cardiovascular profile in shock) of serum lactate more than 2 mmol/L, a decrease in central venous blood saturation of less than 70%, an increase in the arterio-venous carbon dioxide difference of more than 6 mm Hg, and the need for intra-aortic balloon counterpulsation or other extracorporeal methods of circulatory support within 24 hours after surgery.
Regional tissue oxygen saturation levels (rSO2, %) | 24 hours
  Difference between groups in regional kidney near-infrared oximetry (rSO2, %): before sternotomy, at the CPB, 6 hours and 24 hours after surgery.
ΔPCO2/ΔContO2 (ratio) | 24 hours
  Difference between groups in terms of ΔPCO2/ΔContO2: before sternotomy, 6 hours and 24 hours after surgery.
AKI Severity (degree) | 7 days
  Difference between groups in severity of AKI as defined by the KDIGO guidelines:
  Stage 1 AKI is diagnosed when serum creatinine rises 1.5 to 1.9 times its baseline and preoperative values within seven days postoperatively, or when it rises ≥0.3 mg/dL (≥26.5 μm/l) within 48 hours after the intervention, and also if urine output is <0.5 ml/kg/h for 6-12 hours in the first postoperative period.
  Stage 2 AKI is diagnosed when serum creatinine increases 2.0 to 2.9 times its preoperative baseline values within 7 days postoperatively and urine output is <0.5 ml/kg/h more than 12 hours after surgery.
  Stage 3 AKI is diagnosed when serum creatinine rises 3 times its preoperative baseline values within seven days post-intervention, or when it rises to ≥ 4.0 mg/dl (≥ 353.6 μm/L) within 48 hours after the intervention, or if there is a need for renal replacement therapy, and also, if the urine output was <0.3 ml / kg / h within 24 hours after surgery.
AKI duration (hours) | Seven days
  Difference between groups in the duration of AKI: transient (less than 48 hours) and persistent.
Level of NO in exhaled air (ppm) | 1st day after operation
  Difference between groups in the level of NO in exhaled air at baseline, on admission to the ICU, 6 hours later and 24 hours after surgery.
Renal replacement therapy need (%) | 14 days
  Difference between groups in the frequency of need for renal replacement therapy during hospitalization.
Major adverse kidney events (%) | 30 days
  Difference between groups in the frequency of major kidney complications during hospitalization. Major adverse kidney events (MAKE) are a composite endpoint and include death, new episodes of kidney replacement therapy, and deterioration in renal function (GFR decrease of 25% or more from baseline).
Incidence of incomplete recovery of renal function (%) | 30 days
  Difference between groups in the incidence of incomplete recovery of renal function (decrease in GFR by more than 10% compared with preoperative levels), or persistent renal dysfunction (defined as an increase in serum creatinine 1.5 times the baseline values or ≥0.5 mg / dL (44 µmol/L) compared with preoperative level) at discharge from the hospital.
Maximum severity of multiple organ failure (SOFA scale) | 24 hours
  Difference between groups in the level of organ dysfunction and mortality risk measured on a scale Sequential Organ Failure Assessment (SOFA) in the first 24 hours after surgery. Minimum score is 0, maximum score is 24. A higher score indicates an increased risk of mortality.
Vasoactive-inotropic score (VIS) | 24 hours
  Difference between groups in the maximum requirement for inotropic and vasopressor drugs assessed as the vasoactive-inotropic score (VIS). VIS is calculated as follows: dose of dopamine (mcg/kg/min) + dose of dobutamine ( mcg/kg/min) + 100 x dose of epinephrine (mcg/kg/min) + 10 x dose of milrinone (mcg/kg/min) + 10,000 x dose of vasopressin (u/kg/min) + 100 x dose of norepinephrine (mcg /kg/min) + 10 × dose of phenylephrine (mcg/kg/min).
Duration of mechanical ventilation (hours) | 21 days
  Difference between groups in the duration of mechanical ventilation (hours).
ICU stay (days) | 30 days
  Difference between groups in the length of ICU stay (days).
Hospital stay (days) | 30 days
  Difference between groups in the length of hospital stay (days).
Hospital mortality (%) | 14 days
  Difference between groups in hospital mortality rate.
30-day mortality rate (%) | 30 days
  Difference between groups in mortality rate within 30 days after surgery.
Incidence of neurological complications of type 1 (stroke, transient ischemic attack, coma) (%) | 14 days
  Difference between groups in the incidence of neurological complications of type 1 (stroke, transient ischemic attack, coma) during hospitalization.
Incidence of neurological complications of type 2 (delirium, early postoperative cognitive dysfunction, first-onset seizures) (%) | 14 days
  Difference between groups in the incidence of neurological complications of type 2 (delirium, early postoperative cognitive dysfunction, first-onset seizures) during hospitalization.
Platelet count | 24 hours
  Difference between groups in platelet counts 24 hours after surgery.
Postoperative bleeding (mL) | 24 hours
  Difference between groups in the volume of postoperative bleeding, which is calculated as the total blood loss through drains during the stay in the ICU.
Incidence of blood or blood component transfusion (%) | Seven days
  Difference between groups in the frequency of blood transfusion or transfusion of blood components during the period of stay in the ICU.
Incidence of major adverse cardiac events (MACE) (%) | 30 days
  Differences between groups in the incidence of major adverse cardiac events (MACE) during hospitalization and within 30 days after surgery. Major adverse cardiac events - combined endpoint: myocardial infarction, pacing requirement for >48 hours, cardiac arrest.
Incidence of other postoperative complications (%) | 30 days
  Differences between groups in the incidence of other postoperative complications (acute respiratory failure requiring noninvasive ventilation or reintubation, pneumonia, vasoplegia, wound infections, sepsis, readmission to the ICU) to be determined according to standard ESA/ESICM definitions where possible.

OTHER OUTCOMES:
Subclinical AKI | 24 hours
  Differences between groups in the incidence of subclinical AKI according to the results of the study of biomarkers of kidney damage.
Subclinical intestinal injury | 24 hours
  Differences between groups in the incidence of subclinical intestinal injury according to the results of testing the intestinal injury biomarkers.
Subclinical myocardial damage | 24 hours
  Differences between groups in the frequency of subclinical myocardial damage according to the results of the study of biomarkers of myocardial damage.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay O Kamenshchikov, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medic
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.